CLINICAL TRIAL: NCT04141722
Title: AGE-RELATED CHANGES IN SLEEP-DEPENDENT EMOTIONAL MEMORY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Principal Investigator, Rebecca Spencer, Associate Professor, University of Massachusetts, Amherst
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1R56AG058685-01 (NIH)
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Sleep; Age; Emotional Valence
Keywords: Emotional Memory; Memory Consolidation; Age-Related Positivity Effect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep (Experimental)
  Interventions: Behavioral: Overnight sleep
- Wake (Experimental)
  Interventions: Behavioral: Wake

INTERVENTIONS:
Behavioral: Overnight sleep — Participant sent home to sleep overnight wearing PSG.
  Arms: Sleep
Behavioral: Wake — Participant sent to go about normal daily routine, instructed not to nap, drink caffeine, or engage in strenuous exercise.
  Arms: Wake

SUMMARY:
Memory influences emotional well being. Research has shown that having a negative emotional bias contributes to both emotion dysregulation and depression. Conversely, reactivating positive memories has been shown to reduce stress and symptoms of depression. In young adults, sleep is widely implicated in emotional processing, including consolidation of emotional memories. Evidence suggests that aging is associated with changes in emotion, including a positive memory bias and enhanced emotional well-being. These changes have been termed the "age-related positivity effect." However, the influence of sleep on these measures has not been investigated in healthy older individuals. The objective of this research is to understand the role of sleep in emotional memory consolidation and emotional well-being across adulthood. We hypothesize that sleep contributes to the age-related positivity effect in memory and affect. Our alternative hypothesis is that age-related decreases in sleep are responsible for reduced emotional memory processing over healthy aging.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 or 50-80 years of age
* Have no history of a sleep disorder
* Have no history of neurological disease or injury
* Have no history of psychiatric illness (anxiety or mood disorder, schizophrenia, etc.)
* No history of chemotherapy
* Not be taking medications which effect sleep
* Habitually sleep more than 6 or more hours per night
* Be able to walk freely and independently
* Have normal to corrected-to-normal vision

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-12-11 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Memory bias | 12 hr delay between encoding and recognition test
  Corrected recognition of positive versus negative pictures

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Spencer, Principal Investigator — University of Massachusetts, Amherst
Locations (1):
- University of Massachusetts, Amherst, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dalgleish T, Werner-Seidler A. Disruptions in autobiographical memory processing in depression and the emergence of memory therapeutics. Trends Cogn Sci. 2014 Nov;18(11):596-604. doi: 10.1016/j.tics.2014.06.010. Epub 2014 Jul 21. PMID 25060510
- [Background] Ramirez S, Liu X, MacDonald CJ, Moffa A, Zhou J, Redondo RL, Tonegawa S. Activating positive memory engrams suppresses depression-like behaviour. Nature. 2015 Jun 18;522(7556):335-9. doi: 10.1038/nature14514. PMID 26085274
- [Background] Speer ME, Bhanji JP, Delgado MR. Savoring the past: positive memories evoke value representations in the striatum. Neuron. 2014 Nov 19;84(4):847-56. doi: 10.1016/j.neuron.2014.09.028. Epub 2014 Oct 30. PMID 25451197
- [Background] Baran B, Pace-Schott EF, Ericson C, Spencer RM. Processing of emotional reactivity and emotional memory over sleep. J Neurosci. 2012 Jan 18;32(3):1035-42. doi: 10.1523/JNEUROSCI.2532-11.2012. PMID 22262901
- [Background] Jones BJ, Schultz KS, Adams S, Baran B, Spencer RMC. Emotional bias of sleep-dependent processing shifts from negative to positive with aging. Neurobiol Aging. 2016 Sep;45:178-189. doi: 10.1016/j.neurobiolaging.2016.05.019. Epub 2016 May 27. PMID 27459938
- [Background] Leigland LA, Schulz LE, Janowsky JS. Age related changes in emotional memory. Neurobiol Aging. 2004 Sep;25(8):1117-24. doi: 10.1016/j.neurobiolaging.2003.10.015. PMID 15212836
- [Background] Charles ST, Mather M, Carstensen LL. Aging and emotional memory: the forgettable nature of negative images for older adults. J Exp Psychol Gen. 2003 Jun;132(2):310-24. doi: 10.1037/0096-3445.132.2.310. PMID 12825643
- [Background] Mather M, Carstensen LL. Aging and motivated cognition: the positivity effect in attention and memory. Trends Cogn Sci. 2005 Oct;9(10):496-502. doi: 10.1016/j.tics.2005.08.005. PMID 16154382
- [Background] Charles ST, Reynolds CA, Gatz M. Age-related differences and change in positive and negative affect over 23 years. J Pers Soc Psychol. 2001 Jan;80(1):136-51. PMID 11195886
- [Background] Mroczek DK, Kolarz CM. The effect of age on positive and negative affect: a developmental perspective on happiness. J Pers Soc Psychol. 1998 Nov;75(5):1333-49. doi: 10.1037//0022-3514.75.5.1333. PMID 9866191